CLINICAL TRIAL: NCT00018330
Title: Genetics, Metabolism and Weight Loss in Older, Obese Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: AGCG-006-98F
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Obesity
Keywords: Behavioral; Weight Loss; Genetics; Lipoprotein lipase; Visceral fat; Lipoprotein
MeSH Terms: conditions — Obesity; Behavior; Weight Loss

INTERVENTIONS:
Behavioral: Weight Loss

SUMMARY:
This study is designed to determine whether sequence variation in the lipoprotein lipase (LPQ) gene affects the amount of weight loss and metabolic responses during a hypocaloric diet treatment for overweight and obese (BMI=25-35 kg/m2), older (50-65 yrs), sedentary veterans.

DETAILED DESCRIPTION:
Veterans who are 50-65 yrs, non-smoking, sedentary and weight stable with a BMI between 25-35 kg/m2 (120-150% desirable body weight) are recruited and screened via telephone, medical history, and physical exam. Exclusion criteria are: diabetes, hypertriglyceridemia (>400 mg/dl), history of cancer or myocardial infarction, clinical depression, renal, liver or hematologic disease, and medications that affect glucose or lipid metabolism (thiazides, estrogen replacement, beta-blockers). Changes in total and visceral body fat are measured by dual x-ray absorptiometry and computerized tomography, resting energy expenditure and fat oxidation rate by indirect calorimetry, and lipoprotein lipids by enzymatic assay. Glucose tolerance is assessed during a three-hour oral glucose tolerance test with measurement of glucose- and insulin levels every 30 minutes. LPL activity is measured in 3050mg pieces of subcutaneous abdominal and gluteal adipose tissue.

ELIGIBILITY:
* 50-65 yrs, non-smoking, sedentary and weight stable with a BMI between 25-35 kg/m2 (120-150% desirable body weight) are recruited and screened via telephone, medical history, and physical exam.

Exclusion criteria:

* Diabetes,
* Hypertriglyceridemia (>400 mg/dl),
* History of cancer or myocardial infarction,
* Clinical depression,
* Renal, liver or hematologic disease, and
* Medications that affect glucose or lipid metabolism (thiazides, estrogen replacement, beta-blockers).

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 1999-04; Study Completion 2004-03

CONTACTS AND LOCATIONS:
Locations (1):
- VA Maryland Health Care System, Baltimore, Maryland, United States